CLINICAL TRIAL: NCT02089841
Title: Efficacy of Artemether/Lumefantrine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Five Years After Wide Scale Use of the Drug in Tanzania.
Brief Title: Efficacy of Artemether/Lumefantrine for the Treatment of Uncomplicated Malaria.
Acronym: ALE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Richard Mwaiswelo (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Richard Mwaiswelo, Investigator, Muhimbili University of Health and Allied Sciences
Organization: Muhimbili University of Health and Allied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3.0.2011
Record Dates: First submitted 2014-03-15; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Efficacy; Artemether/lumefantrine; Malaria; Children
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artemether/lumefantrine (Experimental): In this single-arm study, patients will be treated with Artemether/lumefantrine, and the first, third and fifth doses of the drug will be given under the direct observation of the health workers. The patients will be followed-up for 42 days, on day 1, 2, 3, 7, 14, 21, 28 and 42 to assess the efficacy of the drug.
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Blood samples will be collected on blood slides and filter papers for asexual parasites assessment both by microscope and molecular genotyping respectively following treatment with artemether-lumefantrine, to assess its efficacy.
  Other Names: Coartem

SUMMARY:
Artemether-lumefantrine has been used in Tanzania as first-line treatment for uncomplicated malaria since 2007. Nonetheless, a report of increased proportion of patients with parasitaemia on day 1 following treatment with artemisinin based combination therapies has emerged from Kenya. Similarly, resistance against artemisinins has been confirmed in South-East Asia and it can spread to Africa. Therefore, the purpose of this study was to assess the efficacy of Artemether-lumefantrine for the treatment of uncomplicated malaria among children after five years of wide scale use of the drug in Tanzania.

DETAILED DESCRIPTION:
Artemisinin based combination therapies (ACTs) are currently recommended by the World Health Organization (WHO) as first-line treatment for uncomplicated malaria in all malaria endemic countries including Tanzania, that adopted the policy in 2007. ACTs have proven to be highly efficacious in different parts of the world with different malaria endemicity. Artemisinins clear asexual parasites rapidly and they are also potent against P. falciparum gametocytes, hence reducing disease transmission and spread of drug resistance. Nonetheless, a report in Kenya shows an increase in proportion of patients with parasitaemia on day 1. Most recently, resistance against artemisinins has been confirmed in four countries of South-East Asia, and it may spread to Africa.

In order to safeguard ACTs life span, WHO recommends all suspected malaria cases to be confirmed with parasitological diagnosis, followed by prompt treatment with effective antimalarials. It also emphasizes on the need to conduct efficacy studies for the first and second line antimalarial treatments after every two years so as to be able to detect resistance early on its course. Therefore, based on this notion, this study aimed to assess the therapeutic efficacy of Artemether/Lumefantrine among children with uncomplicated falciparum malaria in Bagamoyo district, five years after its wide scale use in Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Mono-infection with P. falciparum
* Parasitaemia level of 2000 - 200,000/μL
* Absence of danger signs or signs of severe malaria
* Axillary temperature ≥ 37.5°C or history of fever 24 hours prior to coming to the facility
* Absence of other concomitant infections like pneumonia which can cause fever
* No use of antimalarial drug two weeks prior to the study
* Consent to comply to the protocol.

Exclusion Criteria:

* Presence of general danger signs or signs of severe falciparum malaria
* Severe malnutrition
* Febrile condition due to diseases other than malaria, such as measles, acute lower respiratory infection or other known chronic diseases
* Regular medication which might interfere with antimalarial pharmacokinetics
* History of hypersensitivity reactions or contraindications to any medicine being used in the trial.

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without parasitaemia on day 42. | 42 Days
  Proportion of patients without parasitaemia or with new infection as corrected by molecular genotyping on day 42 will be used to calculate the efficacy of the trial medicine.

SECONDARY OUTCOMES:
Plasma lumefantrine concentration | 7 days and 14 days
  Mean plasma lumefantrine concentration among patients on day 7 and day 14 following treatment with artemether/lumefantrine as a predictor of cure rate.

OTHER OUTCOMES:
Proportional of patients without parasitaemia on day 42 | 42 days
  Proportion of patients without parasitaemia on day 42 as purely assessed by molecular genotyping of all collected samples on this day, differentiate between recrudescence and new infection and use it to calculate the efficacy of the trial medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Martensson, PhD, Study Director — Karolinska Institutet
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania